CLINICAL TRIAL: NCT04187677
Title: Investigation of the Effect of Proprioceptive Sensory Training on Activity Limitation, Functional Use of Hand and Quality of Life in Individuals Undergoing Open Carpal Tunnel Relaxation
Brief Title: Effect of Sensory Training on Activity Limitation, Functional Use of Hand and Quality of Life After Wrist Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Study-1; Halil Ibrahim Ergen (Other: Sanko University)
Record Dates: First submitted 2019-10-21; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Proprioception
Keywords: sensory; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Therapy Group (Active Comparator)
  Interventions: Other: classical hand therapy
- Sensory Training Group (Experimental)
  Interventions: Procedure: Sensory Training

INTERVENTIONS:
Procedure: Sensory Training — The sensory training group includes sensory-oriented interventions and exercises unlike the other classical hand therapy group.
  Arms: Sensory Training Group
Other: classical hand therapy — classical hand therapy
  Arms: Hand Therapy Group

SUMMARY:
The aim of this study is to determine the benefits of sensory training for participants who are included in rehabilitation after carpal tunnel surgery.

ELIGIBILITY:
Inclusion Criteria:

* SANKO University Health Practice and Research Center, Orthopedics and Traumatology Unit underwent open carpal tunnel loosening surgery.

Exclusion Criteria:

* The presence of nerve entrapment other than the median nerve (any sensory / motor deficits in the ulnar or radial nerve),
* Wrist injury history (fractures, carpal instabilities),
* Previous surgery in the hand or wrist region,
* Traumatic and recurrent Carpal Tunnel Syndrome, inflammation of the tendon sheath or the presence of general active inflammation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Joint Position Matching | Baseline (First day)
  In our study, the wrist joint's range of motion will be evaluated in 2 different directions (flexion / extension and radial / ulnar deviation) for proprioception evaluation. For evaluations of all directions, the individual will be required to bring the wrist to the end of the movement, then to perform half the normal range of motion, while the wrist is in a hanging position from the table edge to allow full movement. The difference between the angular value and the angular value created by the individual will be noted by looking at the angular value on the fixed goniometer.
Purdue Pegboard Test | Baseline (First day)
  The Purdue Pegboard Test is a neuropsychological test of manual dexterity and bimanual coordination.
Activity Limitation | Baseline (First day)
  The Patient-Specific Functional Scale is a self-reported, patient-specific outcome measure, designed to assess functional change, primarily in patients presenting with musculoskeletal disorders. The scale was developed by Stratford et al 1995 as a self-report measure of function that could be used in patients with varying levels of independence. It was designed to provide clinicians with a valid, reliable, responsive, and efficient outcome measure that would be easy to use and applicable to a large number of clinical presentations.
Health-Related Quality of Life | Baseline (First day)
  The EuroQoL-five-dimension (EQ-5D) is one of the most commonly used questionnaires to elicit health state utilities, having both a youth and an adult version. For general populations of adults two versions of the questionnaire have been developed, 3L and 5L, with the latter offering a more detailed description of health status. In order to use the EQ-5D to estimate quality-adjusted life-years, a value set to reflect people's preferences for different health states is needed.

CONTACTS AND LOCATIONS:
Locations (1):
- SANKO University, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Derived] Ergen HI, Keskinbicki MV, Oksuz C. The Effect of Proprioceptive Training on Hand Function and Activity Limitation After Open Carpal Tunnel Release Surgery: A Randomized Controlled Study. Arch Phys Med Rehabil. 2024 Apr;105(4):664-672. doi: 10.1016/j.apmr.2023.12.004. Epub 2023 Dec 21. PMID 38142026